CLINICAL TRIAL: NCT01586468
Title: A RANDOMISED, DOUBLE-BLIND, PLACEBO-CONTROLLED PILOT STUDY OF THE EFFICACY AND SAFETY OF WF10 IN SUBJECTS SUFFERING FROM PERSISTENT ALLERGIC RHINITIS
Brief Title: PILOT STUDY OF THE EFFICACY AND SAFETY OF WF10 IN SUBJECTS SUFFERING FROM PERSISTENT ALLERGIC RHINITIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nuvo Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WF10-07-002
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2010-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NaCl Solution (Placebo Comparator)
  Interventions: Drug: NaCl Solution
- WF10 0.5 ml/kg BW (Experimental)
  Interventions: Drug: WF10

INTERVENTIONS:
Drug: WF10 — 0.5 mg/kg B.W.
  Arms: WF10 0.5 ml/kg BW
Drug: NaCl Solution — NaCl Solution
  Arms: NaCl Solution

SUMMARY:
Objectives To assess the efficacy and safety of WF10 infusions in the treatment of subjects with persistent allergic rhinitis.

Study Design Randomized, double-blind, placebo-controlled, parallel-group, single-centre trial.

Subjects 50 subjects (25 per treatment group) with history of persistent allergic rhinitis for at least 2 years prior to enrolment and a positive allergen skin test. Subjects will be required to have a minimum mean score ≥6 for the baseline Total Nasal Symptom Score (TNSS) (mean score of morning and evening reflective TNSS assessments for the 3 days prior to randomization and treatment.

Treatments At the first treatment visit (T1), subjects that comply with the inclusion and exclusion criteria will be randomized into one of two treatment groups: WF10, or placebo.

Each individual treatment dose of study drug solution is 0.5 mL/kg body weight, diluted into 500 mL saline solution. Treatment will be administered once daily for 5 consecutive days (Visits T1-T5) via intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. History of persistent allergic rhinitis for at least 2 years prior to enrolment. Concurrent history of asthma is permitted.
2. Positive allergen skin test to the relevant allergen(s), performed within the previous 2 years prior to enrolment.
3. Mean score ≥6 for the baseline Total Nasal Symptom Score (TNSS)
4. Screening laboratory values within normal range, except those related to the primary disease, including eosinophil count, and elevated glucose is allowed.
5. Age between 18 and 70 years, inclusive.
6. The subject must be able to read and understand German well enough to answer the questions in the TNSS and Mini Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ), without any translation or explanation.
7. If female, the subject:

   1. Cannot become pregnant because she is surgically sterile (hysterectomy or tubal ligation), or is postmenopausal for at least 6 months prior to the screening visit.

      OR
   2. Is not pregnant, with a negative pregnancy test at screening (confirmed at the baseline visit), and uses an acceptable method of contraception with a low failure rate (PEARL Index) (i.e. less than 1% per year) when used consistently and correct (including oral contraceptives, hormone implant, intrauterine device, , male sexual partner(s) surgically sterile, abstinence).
8. Except for persistent allergic rhinitis, the subject is in reasonably good health, as determined by the discretion of the study investigator (based on the physical examination and electrocardiogram [ECG] results).
9. The subject has signed an informed consent form.

Exclusion Criteria:

1. Non-allergic rhinitis, rhinitis medicamentosa, idiopathic rhinitis or sinusitis.
2. History of nasal surgery in the 6 months prior to enrolment.
3. An upper respiratory or sinus infection within the 2 weeks prior to enrolment.
4. Presence of a severely deviated septum, septal perforation, structural nasal defect or large nasal polyps causing obstruction.
5. Use of intramuscular glucocorticosteroids in the 12 weeks prior to enrolment; use of oral, intravenous or medium or high daily dose inhaled glucocorticosteroids (as described in GINA guidelines - see App. III)) in the 4 weeks prior to enrolment; use of topical (nasal or ocular) glucocorticosteroids in the 2 weeks prior to enrolment. .
6. Use of anti-IgE antibodies (e.g. omalizumab) in the 12 weeks prior to enrolment.
7. Use of anti-leukotrienes (e.g. montelukast) in the 4 weeks prior to enrolment.
8. Unwillingness to discontinue prohibited medications and avoid their use during the study (see section 10.1.5 for a complete list of prohibited medications).
9. Severe haematopoetic, cardiovascular, hepatic, renal, neurological or psychiatric disease.
10. Glucose-6-phosphate dehydrogenase deficiency (activity < 60% = < WHO class 4)
11. A female subject who is lactating.
12. Planned travel outside of the study area during the first 22 days of the study.
13. Any infirmity, disability or geographical location that would limit compliance with the protocol.
14. A subject who has previously been randomized into this study, received at least one dose of study treatment and been withdrawn from this trial will not be allowed to re-enter.
15. Use of another investigational drug within the 30 days prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
TNSS | 9 weeks

SECONDARY OUTCOMES:
MiniRQLQ score, POHA score, and rhinometric and spirometric parameters | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gessner, M.D., Principal Investigator — POIS
Locations (1):
- POIS, Leipzig, Saxony, Germany